CLINICAL TRIAL: NCT02646267
Title: The Efficacy and Safety of Dabigatran Etexilate and Different Intensity Warfarin for the Prevention of Stroke and Systemic Embolism in Patients With Non-valvular Atrial Fibrillation
Brief Title: The Efficacy and Safety Study of Dabigatran and Warfarin to Non-valvular Atrial Fibrillation Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SEL102
Record Dates: First submitted 2016-01-03; First posted 2016-01-05 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Dabigatran; Warfarin; Anticoagulation; Elderly
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard intensity warfarin group (Experimental): standard intensity warfarin group， target international normalised ratio(INR) was 2.1-3.0, warfarin baseline dose of 1.25mg daily and then gradually increase the amount to the target INR range(2.1-3.0)
  Interventions: Drug: standard intensity warfarin
- low intensity warfarin group (Experimental): low intensity warfarin group， target international normalised ratio(INR) was 1.7-2.2, warfarin baseline dose of 1.25mg daily and then gradually increase the amount to the target INR range(1.7-2.2)
  Interventions: Drug: low intensity warfarin
- dabigatran etexilate group (Active Comparator): 110mg dabigatran etexilate was administrated twice a day
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: standard intensity warfarin — target international normalised ratio(INR) was 2.1-3.0
  Arms: standard intensity warfarin group
Drug: low intensity warfarin — target international normalised ratio(INR) was 1.7-2.2
  Arms: low intensity warfarin group
Drug: dabigatran etexilate — 110mg, twice a day, oral
  Arms: dabigatran etexilate group

SUMMARY:
The purpose of this trial is to demonstrate the efficacy and safety of dabigatran etexilate and different intensity warfarin for the prevention of stroke and systemic embolism in patients with non-valvular atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of atrial fibrillation
2. Echocardiography confirmed a non-valvular heart disease
3. Age≥60 years

Exclusion Criteria:

1. Unable to cooperate with doctors
2. CHA2DS2-VASc<2
3. Life expectancy of less than 1 year
4. Rheumatic heart disease or dilated cardiomyopathy
5. History of artificial valve replacement surgery
6. Infectious endocarditis
7. Stroke or transient ischemic attack(TIA) within the last 6 months
8. Previous history of intracranial hemorrhage, gastrointestinal, respiratory or urogenital bleeding
9. Previous intolerance/allergy to warfarin or dabigatran etexilate
10. Blood pressure greater than 180/110 mmHg
11. Chronic liver dysfunction, alanine aminotransferase above the normal reference value of the upper limit 3 times
12. Chronic renal failure, serum creatinine clearance rate (Ccr) less than 30 ml / min
13. Patient was receiving antiplatelet or anticoagulant therapy due to other reasons

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
ischaemic stroke | 2 years
  ischaemic stroke was defined as a blockage in an artery that supplies blood to the brain , resulting in a deficiency in blood flow and focal neurological deficit lasting >24 hours.
major haemorrhage | 2 years
  Major haemorrhage was defined as intracranial hemorrhage, gastrointestinal bleeding, bleeding requiring hospitalization and surgical intervention, a reduction of hemoglobin by≥2 g/dL, requiring red blood cells transfusion ≥2 units.

SECONDARY OUTCOMES:
minor bleeding | 2 years
myocardial infarction | 2 years
pulmonary embolism | 2 years
cardiovascular death | 2 years
all-cause mortality | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wu Jun, doctor, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu J, Wang J, Jiang S, Xu J, Di Q, Zhou C, Min X, Pang S, Wang H, Xu D, Guo Y. The efficacy and safety of low intensity warfarin therapy in Chinese elderly atrial fibrillation patients with high CHADS2 risk score. Int J Cardiol. 2013 Sep 10;167(6):3067-8. doi: 10.1016/j.ijcard.2012.11.078. Epub 2012 Nov 28. No abstract available. PMID 23200268